CLINICAL TRIAL: NCT06382350
Title: Glycemic Excursions in Patients With Type 1 Diabetes Mellitus Using Closed-loop Systems (Insulin Pump and Continuous Glucose Monitor) Versus Conventional Treatment in Different Life Situations - an Observational Multicenter Study
Brief Title: Glycemic Excursions in Patients With Type 1 Diabetes Mellitus Using Closed-loop Systems
Acronym: SAFEDRIVE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Jan Broz, Principal Investigator, University Hospital, Motol
Other Study IDs: KHL-002-2024
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Type 1 Diabetes Mellitus; Type 1 Diabetes Mellitus With Hypoglycemia; Drive
Keywords: Type 1 diabetes mellitus; Driving; Closed-loop system
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Study group: Type 1 diabetes patients with insulin pump MiniMed 780 G +CGM (continuous glucose monitoring)
  Interventions: Device: MiniMed 780 G
- Control group: Type 1 diabetes patients with patients treated by multiple daily injections (MDI) + CGM

INTERVENTIONS:
Device: MiniMed 780 G — none, observational study
  Groups: Study group

SUMMARY:
The study aims to compare glycemic excursions during several life situations (such as periods of driving, periods of night sleep, periods of occupation, periods of physical activity, and periods of stress) in patients with type 1 diabetes treated with closed-loop system and multiple daily insulin dose therapy

DETAILED DESCRIPTION:
This national multi-center prospective observational controlled study focuses on the safety of insulin pump closed-loop in patients over 18 with type 1 diabetes while driving. A total of 100 patients (treated with MiniMed 780 G + CGM) will be enrolled in the study group and 20 patients in the control group (treated by multiple daily injections (MDI) + CGM) at 10-20 study centers.

After the inclusion and exclusion criteria evaluation and informed consent signing, each patient receives the Patient Diary. The diary will be used to record the times of observed events during the study period lasting ten days: periods of driving (from-to), periods of night sleep, periods of occupation, periods of physical activity, periods of stress (self-defined), an extra dose of insulin not covered by carbohydrates, an extra dose of carbohydrates not covered by insulin (more variables are required to hide a little bit the primary target of the study).

CGM data obtained during the study period will also be downloaded at the end of the study period.

Finally, the data from the CGM and the patient diary will be compared and analyzed, especially regarding the course of glycemia during driving and the presence of hypoglycemia.

ELIGIBILITY:
Inclusion criteria

Study group:

* type 1 diabetes
* patients aged ≥18 year
* diabetes duration ≥3 years
* regularly driving (non-professional drivers only)
* treated with insulin pump MiniMed 780 G for at least 6 months with closed-loop setting treatment
* willing to fill in the study questionnaires
* signed patient's informed consent form

Control group:

* type 1 diabetes
* patients aged ≥18 years
* diabetes duration ≥3 years
* regularly driving (non-professional drivers only)
* treatment with multiple daily injections (MDI) of insulin therapy and the use of CGM for at least 6 months
* willing to fill in the study questionnaires
* signed patient's informed consent form

Exclusion Criteria (for study and control groups)

* professional drivers
* pregnancy
* inability to be present at the follow-up visit
* inability to complete the study questionnaires
* participation in another clinical study within the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 1 diabetes patients
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The frequency of hypoglycemia during the driving periods | 10 days of CGM measurement
  This outcome evaluates the number of hypoglycemic events (drop of glycemia <3.9 mmol/l) during the driving periods.

SECONDARY OUTCOMES:
Amount of time spent in the glycemic range between 3.9 and 4.5 mmol/l during the driving periods. | 10 days of CGM measurement
  The outcome evaluates the amount of time spent in the glycemic range between 3.9 and 4.5 mmol/l during driving.

OTHER OUTCOMES:
Analysis of glycemia | 10 days of CGM measurement
  This outcome evaluates the mean glycemia and glycemia variability (SD) during the periods of driving and compares them with the same compared with the same variables obtained during the non-driving periods.
Number of alarms generated by the insulin pump | 10 days of CGM measurement
  This outcome assesses the frequency of alarms generated by the insulin pump during preriods of driving and compares them ther same variable generated in non-driving time.
Insulin dosing | 10 days of CGM measurement
  This is to assess the insulin dosing (insulin units/minute) during driving and compare them with the same variable in non-driving time.
Food intake | 10 days of CGM measurement
  This is to assess the food intake (frequency of food intake) while driving and compare them with non-driving time.
Glycemia during the periods of sleep | 10 days of CGM measurement
  The outcome evaluates glycemia (mmol/l) during a night sleep.
Glycemia during the periods of occupation | 10 days of CGM measurement
  The outcome evaluates glycemia (mmol/l) during periods of occupation.
Glycemia during the periods of physical activity | 10 days of CGM measurement
  The outcome evaluates glycemia (mmol/l) during the periods of physical activity.
Glycemia during the periods of stress | 10 days of CGM measurement
  The outcome evaluates glycemia (mmol/l) during the periods of stress.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brož, MUDr., Ph.D., Principal Investigator — Second Medical Faculty, Charles University
Locations (1):
- UH Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No